CLINICAL TRIAL: NCT02477774
Title: Multi-Institutional Randomized Controlled Trial Evaluating Use of Arista Absorbable Surgical Hemostatic Powder in Anterolateral Thigh Donor Sites
Brief Title: Arista for ALT Donor Sites to Reduce Drain Output
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Davol Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ALT Arista
Record Dates: First submitted 2015-06-18; First posted 2015-06-23 (Estimated); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Seroma
Keywords: Anterolateral Thigh
MeSH Terms: conditions — Seroma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arista (Experimental): Arista to ALT donor site
  Interventions: Device: ARISTA
- Control (No Intervention): No Arista to ALT donor site

INTERVENTIONS:
Device: ARISTA — According to the manufacturer, Arista uses Microporous Polysaccharide Hemospheres (MPH) technology to catalyze the clotting cascade and effectively dehydrate tissue to initiate hemostasis in broad areas. Major advantages of Arista are that it has been shown to be safe and effective across multiple surgical disciplines, is completely absorbed in 24-48 hours, and contains no human or animal components
  Arms: Arista

SUMMARY:
This is a single-blinded multi-institutional randomized controlled trial to evaluate the effectiveness of Arista hemostatic matrix powder (Arista® AH, C. R. Bard, Inc. Davol, Warwick, RI) in reducing drainage output in anterolateral thigh (ALT) free flap donor sites. Increased drainage from donor sites can lead to seroma formation with possible secondary infection, delayed hospital discharge, and additional home care needs for drain care. Arista is an inert plant based absorbable surgical hemostatic powder that can be easily applied to broad surgical fields to reduce bleeding and seroma rates. Therefore, its application to free flap donor sites may bear significant potential benefit.

Specific Aim 1: The main hypothesis of the study is that the use of Arista in anterolateral thigh (ALT) free flap donor sites prior to closure will reduce postoperative drain outputs and time to drain removal compared to ALT donor sites closed without Arista.

Specific Aim 2: This study will also evaluate the secondary hypotheses that Arista will reduce postoperative ALT donor site seromas and patient hospital length of stay.

DETAILED DESCRIPTION:
Free tissue transfer is a commonly performed procedure, especially at tertiary care hospitals. In free tissue transfer, "spare tissue" from one area of the body (donor site) is re-implanted to an area that is need of reconstruction (defect site). When relocated, the "spare tissue" is given vitality and blood supply at its new location by microscopically sewing and connecting its feeding artery and vein to an artery and vein in or near the defect site. Hence, this operation is referred to as "microvascular free tissue transfer" or "free flap". Defect sites most commonly result from tumor or cancer removal and trauma related injuries. Free flaps are frequently used to reconstruct breast tissue after mastectomy, head and neck cancer resections, extremity injuries, and chronically infected wounds. The indications, utilization, and expertise in free flap surgery continue to grow, providing patients with enhanced outcomes of otherwise difficult cancers and wounds.

Since its original description in 1984 the ALT microvascular free flap has become an increasingly integral part of head and neck reconstructive surgery.1, 2 ALT free flaps have been shown to be a reliable method for several reconstructive procedures with minimal donor site morbidity.2-4 The ALT free flap is composed of skin, subcutaneous tissue, and fat of the anterolateral thigh. The blood supply to this area is from the lateral circumflex femoral artery and vein. These vessels along with the tissues of the anterolateral thigh are carefully dissected and removed as a single unit to be re-implanted in a different part of the body.

Multiple options exist for soft tissue free flap donor sites similar to the ALT. However, a distinct advantage of the ALT free flap over others is the minimal donor site morbidity that the patient undergoes. Patients are able to fully ambulate and function after the surgery, and are left with only a well-healed scar line. Despite its many advantages, postoperative fluid collections continue to be problematic in the ALT donor site. Studies have reported seroma rates in ALT donor sites as high as 5% although this likely underestimates the true incidence of clinically significant postoperative fluid collections and wound complications in this patient population.2 ALT free flaps require a large amount of tissue dissection and removal, creating a large potential space in the lateral thigh that often requires prolonged postoperative suction drainage and pressure dressings in efforts to minimize fluid accumulation.

Research in optimal postoperative management for the ALT donor site is lacking. Current management without the use of Arista often requires a surgical drain for 7-14 days, which can delay patient discharge and expose patients to increased risk of postoperative wound infections. There is a paucity of data on methods to reduce ALT donor site drain output and seromas. Surgeons often use a combination of closed suction surgical drains and pressure dressings to try and reduce the amount of fluid collection in the thigh donor sites. Although this does provide some advantage, if these techniques are required for a prolonged time, unnecessary hospital stay and patient morbidity are attained. According the Healthcare Cost and Utilization Project, an average inpatient hospitalization in 2009 cost $2,000 per day, and is increasing.5 If the use of a single bottle of Arista could reduce just 1 hospital day per patient it could save at least $80,000 dollars a year at our department alone. Further, the associated morbidity and health care costs of potential seroma or infected seroma complications may be avoided.

A randomized controlled trial aimed at evaluating improved methods to reduce postoperative drainage from ALT donor sites could provide critical information on how to best serve our patients, eliminate unnecessary hospital stay, and reduce overall cost. Once studied in a controlled single flap environment, these methods could be then expanded to other or all free flap donor sites.

According to the manufacturer, Arista uses Microporous Polysaccharide Hemospheres (MPH) technology to catalyze the clotting cascade and effectively dehydrate tissue to initiate hemostasis in broad areas. Major advantages of Arista are that it has been shown to be safe and effective across multiple surgical disciplines, is completely absorbed in 24-48 hours, and contains no human or animal components.6-8

Sindwani et al. was the first to report effectiveness and safety of Arista as a hemostatic agent in otolaryngology demonstrating its application in controlling postoperative bleeding after endoscopic sinus surgery.8 Zhang et al. demonstrated success rate of 100% in the prevention of seromas in patients undergoing resection of malignant tumors in multiple locations, including the lower extremity.7 Arista was recently shown to be useful in reducing postoperative chest tube output and hemostasis time in patients undergoing cardiothoracic surgery.6

These previous works support the idea that Arista could be effective in reducing postoperative fluid collection and drainage time in free flap donor sites. However, this would be a new application of Arista with wide applicability that has not been previously described.

1.1 Research Rationale and Possible Influence On Clinical Practice

Reconstructive surgery has evolved in a recent era of increased attention to patient satisfaction and cost savings. The ALT free flap has been proven to be highly successful; however, optimal management of the donor site postoperatively is an area in need of additional gains via research. Decreasing free flap donor site drain output and earlier drain removal could improve the quality of life of our patients, significantly decrease the cost of their care, and potentially decrease drain-associated infections. If this study were to demonstrate Arista to reduce postoperative donor site drainage and seroma rates and/or a decrease in hospital length of stay resulting from early surgical drain removal, it could dramatically affect the way we take care of our patients.

This study seeks to critically evaluate current clinical practice paradigms to better understand the influence of Arista use in free flap donor sites. A prospective, multi-institutional, randomized, controlled, single-blinded trial is the clearest methodology to evaluate the possible benefits of Arista. Additionally, study in the ALT free flap alone, a single and commonly performed free flap, limits bias and confounding variables. No clinical trial of this level has been performed on this topic; thus, our proposal is novel and the findings of the study are potentially important.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ALT free tissue transfer for head and neck reconstruction
* Patient must be 18 years of age or older.
* The patient must have capacity to be able to sign a study-specific informed consent prior to study entry.

Exclusion Criteria:

* Pregnancy (for female patients).
* Patients who will require anticoagulant medications other than routine DVT prophylaxis within 8 days postoperatively.
* Presence of clotting or bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-07; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Seth, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arista | Control
Started | 29 | 26
Completed | 29 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arista | Control | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (12) | 64 (13) | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 19 | 22 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Drain Output
Description: The primary outcome analyzed in this study will be total drain output (mL) in an effort to determine if the addition of Arista to the wound bed decreases overall wound drainage and drain output.
Time Frame: 1-14 days after Surgery
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Arista | Control
Number analyzed (Participants) | 29 | 26
ml | 284 (153) | 317 (178)

2. Primary Outcome: Number of Participants With the Development of ALT Donor Site Seroma
Description: ALT donor site will be evaluated for seroma
Time Frame: 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Arista | Control
Number analyzed (Participants) | 29 | 26
Participants | 6 | 4

3. Primary Outcome: Timing to Drain Removal
Description: Given that drain output influences time of drain removal, assessment will be made to determine if timing of drain removal differs between groups.
Time Frame: 30 days postoperative
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arista | Control
Number analyzed (Participants) | 29 | 26
days | 5.9 (1.5) | 6.5 (1.6)

4. Secondary Outcome: Hospital Length of Stay
Description: Will eval hospital length of stay for both groups
Time Frame: 30 days postoperative
Population: Hospital Length of Stay data were not collected.
Arm/Group | Arista | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Arista | Control
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26
Other Adverse Events (participants affected / at risk) | 0/29 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT02477774/Prot_SAP_ICF_000.pdf